CLINICAL TRIAL: NCT01163734
Title: A Randomized, Double-blind, Placebo-controlled Study of Ranolazine in Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: Ranolazine in Diastolic Heart Failure
Acronym: RALI-DHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: University Medicine Göttingen, Cardiac Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GS-US-270-0101
Record Dates: First submitted 2010-07-12; First posted 2010-07-16 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2011-03

CONDITIONS: Diastolic Heart Failure
Keywords: Heart Failure with Preserved Ejection Fraction (HFpEF); Coronary Artery Disease (CAD)
MeSH Terms: conditions — Heart Failure, Diastolic; Coronary Artery Disease | interventions — Ranolazine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Experimental)
  Interventions: Drug: Ranolazine
- Saline 0.9% (Placebo Comparator): Saline 0.9% and placebo tablet
  Interventions: Other: Saline 0.9% and placebo tablet

INTERVENTIONS:
Drug: Ranolazine — Intravenous treatment followed oral treatment for 13 days.
  Other Names: Ranexa
  Arms: Ranolazine
Other: Saline 0.9% and placebo tablet — Intravenous treatment followed by oral treatment for 13 days
  Other Names: Normal Saline
  Arms: Saline 0.9%

SUMMARY:
Patients with CAD and clinical symptoms of heart failure or patients with suspected heart failure with preserved ejection fraction (HFpEF) will be enrolled. Study drug will be given as continuous IV infusion followed by oral treatment for 13 days. LV pressures and hemodynamic data will be measured prior to and after administration of study drug. In addition, Doppler ECHO, cardiopulmonary exercise testing (CPET), and NT-pro-BNP determination will be performed. Adverse events and safety labs will be collected and monitored.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled proof-of-concept study of ranolazine in patients with heart failure with preserved ejection fraction (HFpEF). Patients will be randomized to receive ranolazine or placebo in a 1.5:1 ratio (12 ranolazine: 8 placebo).

Treatment will consist of intravenous infusion of study drug followed by oral treatment for a total of 14 days treatment period. Study contact will be made approximately 14 days after the treatment period to assess safety.

Cardiac catheterization will be performed for LV pressures and hemodynamic measurements before and after drug administration. Doppler ECHO, CPET, and NT-pro-BNP determination will be performed at screening and at end of study. Adverse events and safety labs will be monitored and collected.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged > 40 years
2. Clinical symptoms of heart failure (NYHA class II-III) at time of screening (e.g., dyspnea, paroxysmal nocturnal dyspnea, orthopnea, bilateral lower extremity edema)
3. Left ventricular ejection fraction (LVEF) > 45% at screening
4. With:

   * E/E' > 15 measured by Tissue Doppler echocardiography at screening
   * NT-pro-BNP > 220pg/mL at screening
   * Average resting LVEDP >18 mm Hg (refer to continued eligibility criteria),
   * Average resting time constant of relaxation (tau) > 50 ms at time of cardiac catheterization (refer to continued eligibility criteria)
5. Signed informed consent

Exclusion Criteria:

1. Acute cardiac decompensation requiring mechanical ventilation
2. Hypotension with blood pressure < 90/50 mm Hg
3. Primary hypertrophic or restrictive cardiomyopathy or systemic illness associated with infiltrative heart disease (e.g., cardiac amyloidosis)
4. Pericardial constriction
5. Hemodynamically significant uncorrected obstructive or regurgitant valvular disease
6. Cor pulmonale or other causes of right heart failure not associated with left ventricular dysfunction
7. Clinically significant pulmonary disease in the opinion of the Investigator or requiring home oxygen or oral steroid therapy
8. History of serious cardiac dysrrhythmias including atrial fibrillation with resting heart rate of > 100 beats per minute
9. Need for treatment with Class I or III antiarrhythmic medications
10. Implantable pacemaker, cardioverter-defibrillator, or left ventricular assist device
11. Clinically significant chronic hepatic impairment (Child-Pugh Class B [moderate] or Class C [severe])
12. Severe renal insufficiency defined as creatinine clearance ≤30 mL/min as calculated by Cockcroft-Gault formula or Modified Diet in Renal Disease (MDRD) equation.
13. History of congenital or a family history of long QT syndrome, or known acquired QT interval prolongation
14. Inability to exercise due to other co-morbidities that may affect performance of cardiopulmonary exercise test (CPET) (e.g., osteoarthritis, peripheral vascular disease)
15. Current treatment with potent and moderate CYP3A inhibitors
16. Current treatment with potent CYP3A inducers (e.g., rifampin/rifampicin, St. John's Wort, carbamazepin/carbamazepine)
17. Prior treatment with ranolazine
18. Other conditions that in the opinion of the investigator may increase the risk to the patient (e.g. pts with weight ≤60 kg), prevent compliance with study protocol or compromise the quality of the clinical trial

Continued Eligibility Criteria:

Patients must continue to meet eligibility criteria and have an average (of 3 measurements) resting LVEDP > 18 mm Hg and resting tau > 50 ms at time of cardiac catheterization to receive study drug.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 30 minutes in cardiac catheterization hemodynamic parameters at both resting and paced conditions | Baseline to 30 minutes
  Change from baseline to 30 minutes from initiation of study drug bolus No.1 in cardiac catheterization hemodynamic parameters at both resting and paced conditions:
  Time-constant of relaxation (tau)
  Left ventricular end-diastolic pressure (LVEDP)
  dP/dtmin (minimal rate of LV pressure change)

SECONDARY OUTCOMES:
Change from baseline to Day 14 in mitral E wave velocity/mitral annular velocity (E/E') ratio | Baseline to Day 14
Change from baseline to Day 14 in VO2 max | Baseline to Day 14
Change from baseline to Day 14 in N-terminal pro-brain B-type natriuretic peptide (NT-pro-BNP) | Baseline to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Lars S. Maier, MD, Principal Investigator — University Medicine Göttingen, Cardiac Center
Locations (1):
- University Medicine Goettingen (UMG), Göttingen, Germany

REFERENCES:
- [Derived] Maier LS, Layug B, Karwatowska-Prokopczuk E, Belardinelli L, Lee S, Sander J, Lang C, Wachter R, Edelmann F, Hasenfuss G, Jacobshagen C. RAnoLazIne for the treatment of diastolic heart failure in patients with preserved ejection fraction: the RALI-DHF proof-of-concept study. JACC Heart Fail. 2013 Apr;1(2):115-22. doi: 10.1016/j.jchf.2012.12.002. Epub 2013 Apr 1. PMID 24621836
- [Derived] Jacobshagen C, Belardinelli L, Hasenfuss G, Maier LS. Ranolazine for the treatment of heart failure with preserved ejection fraction: background, aims, and design of the RALI-DHF study. Clin Cardiol. 2011 Jul;34(7):426-32. doi: 10.1002/clc.20897. Epub 2011 Apr 27. PMID 21538388